CLINICAL TRIAL: NCT04073134
Title: Cholesterol Reduction With Evolocumab and Coronary MicrovascuLar Function and Coronary Flow: The CHORAL Flow Study
Brief Title: The CHORAL Flow Study
Acronym: CHORAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18HH4626; 2018-002483-11 (EudraCT Number)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Hyperlipidemias
Keywords: Coronary Artery Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Hyperlipidemias | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Randomised control Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Active Comparator): Participants will receive evolocumab 140 mg subcutaneous injections once every 2 weeks.
  Interventions: Biological: Evolocumab
- Placebo (Placebo Comparator): Participants will receive placebo subcutaneous injections once every 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Evolocumab — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen.
  Other Names: Repatha; AMG 145
  Arms: Evolocumab
Drug: Placebo — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen.
  Arms: Placebo

SUMMARY:
CHORAL Flow is a randomised, double blinded, placebo-controlled trial of the effects of evolocumab on coronary flow at 12 weeks.

DETAILED DESCRIPTION:
Evolocumab is a proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor which has been shown in the Fourier Trial to reduce major cardiovascular events in statin-treated patients with raised LDL cholesterol compared to placebo. The precise mechanisms via which evolocumab therapy impacts cardiovascular outcomes remain unknown. Coronary blood flow is a powerful predictor of clinical outcomes across a wide range of cardio-circulatory disorders as well as within normal subjects. Improvement in coronary microvascular function and coronary flow, therefore, could potentially represent one of the core pathways via which evolocumab offers cardiovascular protection. In the CHORAL Flow Study patients will undergo invasive and non-invasive physiological assessment with coronary flow measurements before and after 12 weeks of therapy with evolocumab or placebo. Patients in the treatment arm will go on to have a further non-invasive assessment of coronary flow at 24 weeks of therapy in a single blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18 and 80 years, with a clinical indication for coronary angiography and:

1. willing to provide consent: Provide written (signed and dated) informed consent and be capable of understanding the study and co-operating with treatment and follow-up.
2. raised levels of fasting (>9h) LDL-cholesterol (≥2mmol/L) either on optimal statin therapy (90% of overall sample) or intolerants to statins (restricted to 10% of overall sample). Optimal statin therapy will be defined as at least 4 weeks of atorvastatin 40mg or more, with no change in statin dose during this period.
3. at least one other risk factor for vascular disease or established vascular disease.
4. willing and able to use a highly effective method of contraception from screening until 15 weeks after the last dose of IP if a woman of childbearing potential.

Exclusion Criteria:

1. Patients unable or unwilling to provide written informed consent;
2. Patients unable to undergo cardiac catheterisation;
3. Patients with contraindication to adenosine (severe asthma, second or third degree atrioventricular block, heart rate lower than 40/min at rest, previous formal diagnosis of long QT syndrome, acute decompensated heart failure, severe hypotension, advanced (stage IV) or decompensated chronic obstructive pulmonary disease (COPD);
4. Uncontrolled hypertension (systolic BP >180mmHg or DBP >110mmHg, despite ongoing therapy);
5. Clinical heart failure NYHA class III/IV or Ejection Fraction on imaging modality (Echo, MRI) <40%;
6. Severe valvular heart disease;
7. Severe (>95% diameter) epicardial coronary stenosis;
8. Recent (last 12 months) clinically significant cerebrovascular event (including ischaemic or haemorrhagic events);
9. End-stage renal failure (eGFR < 30 mL/min/1.73m2);
10. Advanced liver disease, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x ULN
11. Current use of PCSK9 inhibitor;
12. Malignancy with life expectancy <1y;
13. Currently or within last 3 months enrolled on another CTIMP;
14. Known allergy to evolocumab or incipients;
15. Women of childbearing potential who are unwilling or unable to use a highly effective method of contraception from screening until 15 weeks after the last dose of IP.
16. Subject is pregnant or breast feeding or planning to become pregnant or to breastfeed during screening, during treatment with IP and/ or within 15 weeks after the end of treatment with IP.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Maximal coronary flow velocity changes from baseline to 12 weeks | Measured at baseline and after 12 weeks of therapy
  Measured invasively using a doppler sensor tipped wire

SECONDARY OUTCOMES:
Coronary Flow Reserve (CFR), measured invasively | Measured at baseline and after 12 weeks of therapy
Hyperaemic Microvascular Resistance, measured invasively | Measured at baseline and after 12 weeks of therapy
Maximal coronary flow (non-invasive) measured non-invasively using ultrasound (echo) | Measured at baseline and after 12 weeks of therapy and in single-blinded extended treatment arm at 24 weeks
Coronary Flow Reserve (CFR) (Non-invasive) measured non-invasively using ultrasound (echo) | Measured at baseline and after 12 weeks of therapy and in single-blinded extended treatment arm at 24 weeks

OTHER OUTCOMES:
Coronary wave intensity analysis derived from invasive pressure and flow measurements | Measured at baseline and after 12 weeks of therapy
  Exploratory outcome
Exercise coronary flow reserve (CFR) (Non-invasive) measured non-invasively using ultrasound (echo). | Measured at baseline and after 12 weeks of therapy and in single-blinded extended treatment arm at 24 weeks
  Exploratory outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Petraco, PhD, Principal Investigator — Imperial College London; Henry Seligman, MBBS, Study Director — Imperial College London
Locations (1):
- Imperial College NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No